CLINICAL TRIAL: NCT07364708
Title: Effect of Anterior Chamber Deflation Before Reduction of a Detached Descemet's Membrane
Brief Title: AC Deflation in Descemet's Membrane Detachment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Khalafallah, lecturer of ophthalmology, faculty of medicine, Minia university, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 592\7\2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-07

CONDITIONS: Descemet's Membrane Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- will undergo direct intracameral air injection (Other)
  Interventions: Procedure: group A will undergo direct intracameral air injection and group B will undergo anterior chamber deflation then intracameral air injection
- will undergo anterior chamber deflation then intracameral air injection (Other)
  Interventions: Procedure: group A will undergo direct intracameral air injection and group B will undergo anterior chamber deflation then intracameral air injection

INTERVENTIONS:
Procedure: group A will undergo direct intracameral air injection and group B will undergo anterior chamber deflation then intracameral air injection — a group will undergo direct intracameral air injection and another group will undergo anterior chamber deflation then intracameral air injection

SUMMARY:
using a relatively new technique to manage post-cataract surgery complication and measuring its efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patients with post cataract surgery DM detachment diagnosed within 1st week postoperatively.
* Patient age ranges from 50 to 70 years old.

Exclusion Criteria:

* Less than one third of Descemet's Membrane is included.
* Post-operative infection or severe inflammation.
* Patient with pre-existing glaucoma.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of complete anatomical reduction of DMD on ASOCT at the 1-week visit. | 1 week

SECONDARY OUTCOMES:
. Time to complete anatomical reduction (days) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Khalafallah, Minya, None Selected, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol